CLINICAL TRIAL: NCT04327921
Title: A Peer Navigator Model to Improve Quit Attempts and Smoking Cessation Rates Among HIV-positive Smokers
Acronym: P-NAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Patricia Cioe, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21CA243906-01 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-31 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: HIV
Keywords: HIV; HIV Virus; smoking; smoking cessation; peer navigator; social support; self efficacy; quit smoking; smoking treatment; quitting smoking
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Once the baseline interview is complete, the principal investigator, who is not involved in conducting assessments, will randomize eligible participants to one of two study conditions. Urn randomization will be used to ensure the groups are balanced on gender and Fagerström Test of Nicotine Dependence (FTND) score. The Research Assistant will not be informed of treatment condition assignment. All participants will be scheduled for a week 1 session with a study nurse within one week of the baseline appointment. The nurse will use a detailed counseling manual to ensure standardization of treatment delivery.
Who Masked: Outcomes Assessor
Masking Description: The research assistant will not be aware of study condition of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peer navigation social support for smoking cessation (Experimental): 36 HIV-positive smokers will have a 30-minute session with the study nurse to discuss smoking cessation. They will also discuss the importance of social support for quitting and the role of a Peer Navigator. Those participants who set a quit date will choose medication/s in collaboration with the nurse and/or physician. The Peer Navigator will be introduced and will reinforce adherence to medication. The Peer Navigator will ensure that the patient picks up the medication, and will help to manage side effects via physician/nurse consultation. The Peer Navigator will provide social support for quitting via weekly phone calls for 12 weeks.
  Interventions: Behavioral: Peer navigation social support for smoking cessation
- Standard Condition (Active Comparator): 36 HIV-positive smokers will receive standard care. Participants will meet for a 30-minute session with a study nurse. They will receive counseling based on the 5A's. The nurse will ask about current smoking habits, advise the participant to quit, assess readiness to quit, and assist by providing resources (community programs, Quit line phone number). The nurse will calculate Lung Age which will serve as a motivation tool to encourage smokers to quit. Those willing to set a quit date will be instructed to call their physician for cessation medication and will provided with the National Cancer Institute self-help pamphlet. Those participants not willing to set a quit date will be instructed to contact their physician when they are ready.
  Interventions: Behavioral: Standard Condition

INTERVENTIONS:
Behavioral: Peer navigation social support for smoking cessation — Standard guidelines will be used for brief advice for smoking cessation based on the 5A's. Also, motivational interviewing/guidance will also be used to determine whether enhanced treatment (using a Peer Navigator to navigate smoking cessation, obtain medication and treatment, improve adherence to treatment, and provide social support for quitting) will increase participant's quit attempts and smoking cessation rates.
  Arms: peer navigation social support for smoking cessation
Behavioral: Standard Condition — Standard guidelines will be used for brief advice for smoking cessation based on the 5A's.
  Arms: Standard Condition

SUMMARY:
Effective antiretroviral therapy has led to an increased lifespan for persons living with HIV (PLWH), when diagnosed early and engaged in care. This transition to HIV as a chronic illness has resulted in cancer being a leading cause of morbidity and mortality in PLWH. The increased risk of cancer is due in part to a high prevalence of risk factors for cancer - most notably tobacco use. Smoking prevalence is substantially higher in PLWH (40%) compared with the general population (15%) and is associated with increased rates of lung cancers, and other malignancies. Furthermore, combined data from three national surveys showed that the proportion of deaths attributed to AIDS-defining cancers decreased from 2000 to 2010, while the proportion of deaths attributed to non-AIDS-related cancers increased significantly over the same period of time. Smoking cessation studies in PLWH have demonstrated disappointing outcomes, with low quit rates, poor adherence to therapy, and a lack of sustained abstinence. In an HIV and smoking review, it was suggested that research develop focused interventions that targets: 1) adherence to smoking cessation medications, 2) self-confidence for quitting, and 3) social support for smoking cessation. The investigators are proposing is specifically designed to address these 3 targets by using peer navigators to facilitate access to effective smoking treatments and to support abstinence. This study is highly innovative in its application of peer navigators to improve HIV-positive smokers' access to and utilization of existing resources to improve smoking cessation outcomes. The proposed study will provide initial evidence of whether targeting mechanisms of behavior change (self-efficacy and social support) during a quit attempt using peer navigators is effective at improving outcomes. If demonstrated to be successful, it has significant implications for the transformation of current clinical approaches to smoking cessation in HIV clinics. This approach could then be widely implemented to improve outcomes in this group of smokers.

DETAILED DESCRIPTION:
Aims - The specific aims are to examine: (1) the feasibility, acceptability, and initial efficacy of Peer Navigation for Social Support - Smoking in a 24-week randomized pilot study; (2) to compare the effect of Peer Navigation for Social Support, relative to standard care, on mechanisms thought to underlie smoking abstinence in HIV-positive smokers.

Methodology - The investigators will adapt an existing, highly effective peer navigation training program to increase engagement in care within the HIV clinic. The peer navigator for smoking cessation will be a former daily smoker who quit smoking 1-2 years ago and has remained smoke-free. The investigators will train the peer navigator, enroll 6 HIV-positive smokers to test the intervention, and finalize the protocol. The investigators will refine the protocol based on feedback from the peer navigator, the 6 participants, and the study nurses. Next, the investigators will conduct a pilot randomized trial (N = 72) to test the feasibility, acceptability, and initial efficacy of peer navigation in a randomized, 2-group, repeated measures design. The investigators will randomize 36 HIV-positive smokers to each condition: Peer Navigation or standard care. Assessments will be collected at baseline, and at 4-, 12-, and 24-weeks.

Participant Population - Participants for this study will include 78 participants recruited from Providence, Rhode Island.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with HIV
* at least 18 years of age
* smoke at least 5 cigarettes per day for longer than one year
* have an exhaled carbon monoxide (CO) level greater than 5 at baseline

Exclusion Criteria:

* currently using pharmacotherapy for smoking cessation
* an unstable medical or psychiatric condition (defined as a medical or psychiatric hospitalization in the 30 days prior to enrollment)
* experiencing psychotic symptoms
* past-month suicidal ideation or past-year suicide attempt
* pregnant or nursing
* Blood pressure reading greater than 160/100
* Heart Rate less than 45 or greater than 115
* family/household member already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability | Week 24
  Session attendance (recorded as a continuous variable ranging from 1 to 4 study sessions).
Quit Attempts | Week 24
  A quit attempt is defined as a period of 24 hours of no cigarette smoking
Point prevalence abstinence | Week 24
  Biochemically verified 7-day point-prevalence abstinence. Point-prevalence abstinence will be verified by saliva cotinine radioimmune assay analysis (cutoff value of < 15 ng/ml) for stated abstinence of 7 days or longer in those not currently using NRT or other nicotine-containing products. Self-report will always be overridden by objective verification of abstinence in the final analyses. Breath samples for CO will be obtained at each study visit.
Treatment Satisfaction | Week 24
  CSQ-8 will be used to compare treatment satisfaction by study condition.

SECONDARY OUTCOMES:
Change in social support for quitting from baseline to week 12 | Week 12
  Assessed using the Partner Interaction Questionnaire, which assesses negative and positive support for quitting. Participants will be instructed to include all forms of support for quitting (including PN support if assigned to the PNSS-S condition).
Change in self-efficacy for smoking cessation from baseline to week 12 | Week 12
  Contemplation Ladder, a one-item Likert-type scale (rating 1-10). In participants who set a quit date, adherence to pharmacotherapy will be measured via participant self-report and pharmacy refill report at each study session.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Cioe, PhD, Principal Investigator — Brown University
Locations (1):
- Miriam Immunology Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Cioe PA, Pinkston M, Stang GS, Tashima KT, Kahler CW. Peer Navigation for Smoking Cessation in People With HIV Who Smoke: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2025 Feb 24;27(3):517-524. doi: 10.1093/ntr/ntae214. PMID 39251402

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04327921/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04327921/ICF_001.pdf